CLINICAL TRIAL: NCT06126731
Title: PROMIZE: A Phase I/II Trial to Assess the Safety, Tolerability and Preliminary Anti-tumour Activity of Oral Combination Antibiotic Therapy to Modulate the Microbiome in Combination With Enzalutamide With Metastatic Castration Resistant Prostate Cancer (mCRPC).
Brief Title: Combination Study of Antibiotics With Enzalutamide (PROMIZE)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Prostate Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCR5461
Record Dates: First submitted 2023-10-25; First posted 2023-11-13 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Keywords: Microbiome; Antibiotic; Enzalutamide
MeSH Terms: interventions — enzalutamide; Amoxicillin; Metronidazole; Vancomycin; Ciprofloxacin

STUDY DESIGN:
Intervention Model Description: Patients with histologically or cytologically confirmed mCRPC who have previously progressed on at least one line of taxane chemotherapy (or not fit or not willing to receive a taxane) and a next generation antiandrogen (e.g. enzalutamide, apalutamide, darolutamide, abiraterone acetate)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- mCRPC patients dose with a combination of enzalutamide and antibiotics (Experimental): Phase I:
  The evaluation of the safety and tolerability of the combinations of amoxicillin plus metronidazole, and ciprofloxacin plus vancomycin with enzalutamide.
  Phase II:
  Determination of the anti-tumour activity of the combinations of amoxicillin plus metronidazole, and ciprofloxacin plus vancomycin with enzalutamide.
  Interventions: Drug: Enzalutamide 40mg; Drug: Amoxicillin 500mg; Drug: Metronidazole 400mg; Drug: Vancomycin 125mg; Drug: Ciprofloxacin 500g

INTERVENTIONS:
Drug: Enzalutamide 40mg — Enzalutamide is presented in 40mg yellow film-coated tablets. They are supplied in a cardboard wallet incorporated a PVC/PCTFE/aluminium blister pack which holds 28 tablets. Each carton contains 4 wallets (112 tablets in total)
  Other Names: Xtandi
Drug: Amoxicillin 500mg — Red / Buff coloured size '0' capsules containing white to off white powder printed with 'AMOXY 500 ' in black ink
  OR
  White to off-white granular powder filled in hard gelatine capsule shells size '0'. Scarlet colour cap, buff colour body printed with 'AMOXY' on cap and '500' on body
  OR
  White/Maroon size '0' capsules containing white to yellowish granular powder
Drug: Metronidazole 400mg — Yellow, circular (11mm), biconvex, film-coated tablets with '400' debossed on one side and plain on other side
  OR
  White to off white coloured, caplet shaped (17.00 x 6.00 mm) film-coated tablets, debossed "400" on one side and plain on other side
  OR
  Off-white coloured, round, biconvex uncoated tablets engraved "MZ 400" & break line on one side and plain on other
Drug: Vancomycin 125mg — Grey/pink 17.8 ± 0.40 mm hard capsules each containing 125mg, containing white to off white congealed liquid mixture as solid mass
  OR
  Dark blue and brown hard capsules, imprinted with 3125 in red ink
  OR
  Brown 21.4 ± 0.40 mm hard capsule, containing white to off white congealed liquid mixture as solid mass
Drug: Ciprofloxacin 500g — White to off white, capsule shaped, film coated tablets, with a score line on one side and debossed with 'F22' on the other side. The tablet can be divided into equal doses. The size is 18.2 mm x 8.1 mm
  OR
  White, caplet shaped film-coated tablets debossed with '500' on one side and plain on the other side
  OR
  White to off-white, capsule shape, biconvex with bevelled edge, film coated tablet with inscription 'CI' on one side and plain on the other side
  OR
  White, oval shaped film-coated tablets debossed 'C500' on one side and breakline on other side

SUMMARY:
PROMIZE is an open-label, multi-centre, single-arm, Phase I/II clinical trial, evaluating the safety, tolerability and anti-tumuor efficacy of an antibiotic combination and enzalutamide in patients with metastatic castration-resistant prostate cancer (mCRPC).

DETAILED DESCRIPTION:
Patients with histologically confirmed metastatic castration-resistant adenocarcinoma of the prostate refractory to conventional therapy (or for which no conventional therapy exists or is declined by the patient), that have progressed after at least 1 line of taxane based chemotherapy (or not fit or not willing to receive a taxane) and a NAAT are eligible for the study. The Phase I will evaluate the safety and tolerability of the combination of amoxicillin plus metronidazole (2 weeks) followed by ciprofloxacin plus vancomycin (2 weeks) administered for 2 cycles (i.e., 8 weeks) in addition to enzalutamide (160 mg daily). Enzalutamide will continue beyond the completion of the antibiotic combination until disease progression, intolerance, or withdrawal from the study. The DLT period is 4 weeks and commences at the time of combination treatment with antibiotics plus enzalutamide. Each cycle of treatment will be 4 weeks in length.

The design permits the safety monitoring of DLT regularly throughout the 2 phases. During the Phase I study, if 2 or more patients experience a DLT out of up to 6 patients, the schedule will be deemed intolerable, and a decision will be made by the SRC to modify the schedule depending on the timing and nature of toxicity observed and its causality. For any modified schedule, a further 6 patients will be treated, and the new dose and schedule will only be deemed tolerable if no more than 1 out of 6 patients experience a DLT.

The Phase II study will employ a 2-stage design. It will recruit a maximum of 33 patients with a desirable response level of 30% and an undesirable response rate of 10%. Patients enrolled to the Phase I who are treated at the RP2D and are evaluable for response will contribute to the Phase II study. Patients will receive the same dose and schedule deemed to be safe in the Phase I.

In the phase II study, the first stage will enrol 15 patients who are evaluable for response. If at least one patient responds during stage 1, a further 18 patients will be recruited (stage 2). The decision to proceed to stage 2 can be made once one response has been observed after thorough review of the cases where objective response was observed by the SRC. The trial will be terminated with the conclusion that the treatment is futile if no responses are observed in the first 15 patients. The second stage of the trial will enrol 18 patients who are evaluable for response. If >6 patients respond across the 2 stages, the study will have met its efficacy threshold. Further details of the Simon 2-stage design are specified in section 13. If <7 patients respond across the 2 stages, all samples will be analysed to identify predictive biomarkers of response. If a robust biomarker is identified, the study may be expanded in a biomarker-selected cohort following protocol amendment. Further safety analysis of safety (at least 2 further interim looks) will occur throughout the phase II trial.

Approximately 6 patients will be enrolled to the Phase I and up to a total of 33 response evaluable patients will be enrolled to the Phase II study. Patients in the Phase I study who are treated with the RP2D and are evaluable for response can contribute to the Phase II study. Based on this, up to 39 response evaluable patients will be recruited across the 2 phases. Based on a recruitment rate of 3 patients per month across the 2 sites, recruitment will be completed within 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically proven metastatic castration-resistant prostate cancer or adenocarcinoma refractory to conventional treatment, or for which no conventional therapy exists or is declined by the patient.
2. Documented prostate cancer progression as assessed by the investigator with RECIST (v1.1) and PCWG3 criteria with at least one of the following criteria:

   1. Progression of soft tissue/visceral disease by RECIST (v1.1) and/or,
   2. Progression of bone disease by PCWG3 bone scan criteria and/or,
   3. Progression of PSA by PCWG3 PSA criteria and/or
   4. Clinical progression with worsening pain and need for palliative radiotherapy for bone metastases.
3. Phase I: Patients that have progressed after at least 12 weeks of treatment with a NAAT within the previous 6 months Phase II: Patients that have progressed after at least 12 weeks of treatment with a NAAT within the previous 6 months (for combination treatment) or more than 6 months prior to trial entry (for enzalutamide alone resistance run-in).
4. Previously progressed on at least one line of taxane chemotherapy (or not fit or not willing to receive a taxane).
5. Ongoing androgen deprivation maintaining serum testosterone of less than 50 ng/dL (less than 2.0 nM) is mandatory.
6. Life expectancy of at least 12-weeks.
7. Able to swallow tablets.
8. Archival tumour tissue must be available for analyses.
9. Willing to have pre- and post-treatment biopsies if biopsy is feasible.
10. World Health Organisation (WHO) performance status of 0-2 (Appendix 1).
11. Haematological and biochemical indices within the ranges shown below. These measurements must be performed within one week (Day -7 to Day 1) prior to the patient's first dose of IMP.

    Haemoglobin (Hb): ≥ 9.0 g/dL

    Absolute neutrophil count: ≥ 1.5 x 109/L

    Platelet count: ≥ 75 x 109/L

    Serum bilirubin: ≤ 1.5 x upper limit of normal (ULN)

    Alanine aminotransferase (ALT): ≤ 2.5 x (ULN) unless raised due to tumour in which case up to 5 x ULN is permissible

    Aspartate aminotransferase (AST): ≤ 2.5 x (ULN) unless raised due to tumour in which case up to 5 x ULN is permissible

    Serum creatinine / calculated creatinine clearance: ≤ 1.5 x upper limit of normal (ULN) / GFR ≥ 50 mL/min (uncorrected value)

    Serum albumin: >25 g/L
12. 18 years or over
13. Written (signed and dated) informed consent and be capable of co-operating with treatment and follow-up
14. Willing and able to comply with the study requirement including the collection of blood, fresh tumour biopsy, urine, rectal swab and stool samples.

Exclusion criteria:

1. Surgery, radiotherapy, chemotherapy, or other anti-cancer therapy within 4-weeks prior to trial entry into the study (6 weeks for bicalutamide). The use of bisphosphonates or RANK ligand inhibitors in patients with known osteopenia or osteoporosis or bone metastases is permitted. Prior antiandrogenic treatment exclusions as follows:

   * Patients receiving enzalutamide immediately preceding the trial will be able to continue on enzalutamide without washout.
   * Prior flutamide treatment during previous 4-weeks. N.B. Patients whose PSA did not decline in response to antiandrogens given as a second line or later intervention will only require a 14-day washout;
   * Prior bicalutamide (Casodex) and nilutimide (Nilandron) treatment during previous 6-weeks;
   * Prior progesterone, medroxyprogesterone, progestins, cyproterone acetate, tamoxifen, and 5-alpha reductase inhibitors during previous 2-weeks (14-days).
2. Ongoing toxic manifestations of previous treatments. Exceptions to this are alopecia or certain Grade 1 toxicities, which in the opinion of the Investigator and the DDU should not exclude the patient.
3. Previous treatment with any systemic antibiotic within 12 weeks of study entry.
4. Known hypersensitivity reaction or intolerance to any penicillin, amoxicillin, metronidazole, vancomycin, ciprofloxacin or enzalutamide.
5. History of tendon disorder secondary to quinolones
6. Use of drugs that are listed in the prohibited concomitant medications section including strong inducers and inhibitors of CYP450 (please refer to http://medicine.iupui.edu/clinpharm/ddis/table.aspx). Seville orange or grapefruit products and any herbal medications should be avoided for 4 weeks prior to starting trial treatment.
7. Concurrent treatment with prohibited medications which include medications that causes ototoxicity, neurotoxicity, and nephrotoxicity.
8. Known or suspected leptomeningeal metastases or untreated brain metastasis. Patients with brain metastases that have been treated and have been shown to be radiologically stable for more than 6 months may be considered for the trial.
9. History of stroke, epilepsy or current excessive alcohol intake. History of clinically significant hearing loss including but not limited to congenital hearing loss, need for hearing aids, ongoing acute or chronic ear infection, history of tympanic membrane perforation, tinnitus, vertigo, Meniere disease, cerebrovascular ischemia.
10. History of clinically significant hearing loss including but not limited to congenital hearing loss, need for hearing aids, ongoing acute or chronic ear infection, history of tympanic membrane perforation, tinnitus, vertigo, Meniere disease, cerebrovascular ischemia.
11. Patients with partners of child-bearing potential (unless they agree to use a barrier method of contraception [condom plus spermicide] or to sexual abstinence effective from the first administration of any of the investigational agents, throughout the trial and for 6 months afterwards. Patients with partners of child-bearing potential must also be willing to ensure that their partner uses an effective method of contraception for the same duration for example, hormonal contraception, intrauterine device, diaphragm with spermicidal gel or sexual abstinence). Patients with pregnant or lactating partners must be advised to use barrier method contraception (for example, condom plus spermicidal gel) to prevent exposure of the foetus or neonate.

    NB. Abstinence is only considered to be an acceptable method of contraception when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
12. Any condition that would increase enteral absorption in the opinion of the investigator, including but not limited to malabsorption syndromes, impaired GI motility, chronic pancreatitis, partial or complete gastric and/or bowel resections, history of clinically significant gastrointestinal bleeding in the last 6 months, history of mesenteric ischemia or bowel obstruction, chronic diarrhoea (≥Grade 2), inflammatory bowel disease (Crohn's disease, ulcerative colitis).
13. At high medical risk because of non-malignant systemic disease including active uncontrolled infection.
14. Clinically significant history of liver disease consistent with Child-Pugh Class B or C, including viral or other hepatitis, current alcohol abuse, or cirrhosis.
15. Known to be serologically positive for hepatitis B, hepatitis C or human immunodeficiency virus (HIV).
16. Any of the following cardiac criteria:

    * Clinically important abnormalities including rhythm, conduction or ECG changes (left bundle branch block, third degree heart block).
    * Factors predisposing to QT prolongation including congenital long QT syndrome; family history of prolonged QT syndrome, unexplained sudden death (under 40); concomitant medications known to prolong QT interval.
    * Concurrent congestive heart failure, prior history of class III/ IV cardiac disease (New York Heart Association [NYHA] - refer to Appendix 5), prior history of cardiac ischaemia or prior history of cardiac arrhythmia.
    * QTcF (corrected using Fredericia formula) of ≥460 ms.
17. Prior bone marrow transplant or have had extensive radiotherapy to greater than 25% of bone marrow within eight weeks.
18. Active or uncontrolled autoimmune disease requiring corticosteroid therapy or other forms of systemic immunosuppression.
19. Patient is a participant or plans to participate in another interventional clinical trial, whilst taking part in this study. Participation in an observational trial would be acceptable.
20. Any other condition which in the Investigator's opinion would not make the patient a good candidate for the clinical trial.
21. Malignancy other than prostate cancer within 3-years of trial entry with the exception of adequately treated basal cell carcinoma. Cancer survivors, who have undergone potentially curative therapy for a prior malignancy must have no evidence of that disease for at least-3 years and be deemed at negligible risk for recurrence, are deemed eligible.
22. Symptoms of COVID-19 and/or current documented COVID-19 infection.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 39 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Confirm the safety and tolerability of the combination of amoxicillin plus metronidazole (2 weeks) followed by ciprofloxacin plus vancomycin (2 weeks) along with enzalutamide in Phase I in mCRPC patients. | 28 days
  Determine a dose at which no more than one patient out of up to 6 patients experiences a highly probable or probably drug-related DLT, during the 28-day DLT period.
Describe the safety profile of the antibiotic combinations along with enzalutamide in Phase I. | 28 days
  Causality and grading severity of each adverse event related to the investigational agents according to the NCI CTCAE v5.0.
Determine the response rate of the antibiotic combinations in patients with mCRPC in Phase II. | 28 days
  Anti-tumour activity will be defined by response rate on the basis of the following outcomes. If any of the following occur, patients will be considered to have responded:
  * PSA decline ≥ 50% criteria confirmed 4 weeks or later, and/or
  * Confirmed soft tissue objective response by RECIST (v1.1) in patients with measurable disease.

SECONDARY OUTCOMES:
To document possible anti-tumour activity in patients in Phase I. | 28 days
  Antitumour activity will be defined by response rate on the same basis as that used for the primary objective of the Phase II component.
To evaluate progression-free survival (PFS) in mCRPC patients receiving the antibiotic combinations in Phase I. | 12 months
  PFS will be measured from the date of antibiotic commencement to the date of progression as determined by radiological criteria (RECIST v 1.1, PCWG3 bone scan criteria) or unequivocal clinical progression necessitating drug discontinuation (e.g. worsening pain, spinal cord compression, need for other anticancer therapy).
To evaluate PFS in mCRPC patients receiving the antibiotic combinations along with enzalutamide in Phase II. | 12 months
  PFS will be measured from the date of antibiotic commencement to:
  * The date of progression as determined by radiological criteria (RECIST v1.1, PCWG3 bone scan criteria) and/or
  * Unequivocal clinical progression necessitating drug discontinuation (e.g. worsening pain, spinal cord compression, need for other anticancer therapy).
To determine the time to PSA progression from the date of antibiotic commencement | 28 days
  This is an estimate of the biochemical anti-tumour activity of the combination of amoxicillin plus metronidazole (2-weeks) followed by ciprofloxacin plus vancomycin (2-weeks) along with enzalutamide.
To determine the duration of PSA decline as an estimate of the biochemical anti-tumour activity of the combination of amoxicillin plus metronidazole (2-weeks) followed by ciprofloxacin plus vancomycin (2-weeks) along with enzalutamide. | 28 days
  The duration of PSA decline by ≥ 50% is an estimate of the biochemical anti-tumour activity of the combination of amoxicillin plus metronidazole (2-weeks) followed by ciprofloxacin plus vancomycin (2-weeks) along with enzalutamide.
To determine the maximum percentage and absolute PSA decline from baseline | 28 days
  This is an estimate of the biochemical anti-tumour activity of the combination of amoxicillin plus metronidazole (2-weeks) followed by ciprofloxacin plus vancomycin (2-weeks) along with enzalutamide.
To determine the radiologic PFS (rPFS) of the combination of antibiotics and enzalutamide in Phase II. | 12 months
  Radiologic PFS (rPFS) measured from the date of of antibiotic commencement to:
  * Progression of soft tissue/visceral disease by RECIST (v1.1) and/or,
  * Progression of bone disease by PCWG3 bone scan criteria
  * And/or death from any cause
To determine the time to radiologic progression to the combination of antibiotics and enzalutamide in Phase II. | 28 days
  Time to radiologic progression defined from the date of antibiotic commencement to radiologic progression by RECIST v1.1 and/or PCWG3 criteria.
To estimate the OS in mCRPC patients receiving the antibiotic combinations along with enzalutamide in Phase II. | 28 days
  OS will be measured from the date of antibiotic commencement to date of death (whatever the cause).
To further characterise the safety and tolerability profile of the antibiotic combinations with enzalutamide in Phase II. | 28 days
  Causality and grading severity of each adverse event related the investigational agents according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 (v5.0)
To identify biomarkers of response to the antibiotic combinations and of anti-tumour activity in Phase II. | 28 days
  Biomarkers of response include tumour genomics and immunologic characteristics in tumour biopsies from responders and non-responders
To evaluate the peripheral circulation neutrophil-to-lymphocyte ratio (NLR) as a determinant of response to to treatment in Phase II. | 28 days
  NLR at baseline and on-treatment for:
  * Baseline NLR as a determinant of response
  * Percentage change in NLR between baseline and NLR nadir between responders versus non-responders

OTHER OUTCOMES:
To report the effect of the antibiotic combinations on the circulating immune cell repertoire. | 28 days
  Serial peripheral white blood cell immunophenotyping.
To report the effect of the antibiotic combinations on the tumour. | 28 days
  Tumour cytokine analyses
To report the effect of the antibiotic combinations on the circulating chemokine and cytokine expression. | 28 days
  Whole blood cytokine analyses by ELISA.
To evaluate the impact of the antibiotic combinations on whole blood transcriptomes. | 28 days
  Serial whole blood transcriptome analyses.
To evaluate the impact of the antibiotic combinations on tumour genomic evolution. | 28 days
  Serial circulating cell free DNA (cfDNA)

CONTACTS AND LOCATIONS:
Overall Officials: Johann De Bono, MD, Principal Investigator — National Health Service, United Kingdom
Locations (2):
- Oncolgy Institute of Southern Switzerland (IOSI), Bellinzona, Switzerland
- The Royal Marsden NHS Foundation Trust, Sutton, United Kingdom